CLINICAL TRIAL: NCT02135653
Title: A Feasibility Study Followed By A Randomized Phase II Study Of Yoga For Radiation Therapy Side Effects In Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 05813
Record Dates: First submitted 2014-05-02; First posted 2014-05-12 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Feasibility Phase: Eischens Yoga Group
  Interventions: Radiation: Radiotherapy; Other: Eischens Yoga
- Phase II: Eischens Yoga Group
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy
Other: Eischens Yoga
  Groups: Feasibility Phase: Eischens Yoga Group

SUMMARY:
This study will ascertain the feasibility and effect of Eischens yoga interventions on radiation related fatigue, sexual dysfunction and urinary incontinence in stage I /II prostate cancer patients undergoing radiotherapy with photons and/or protons without prostatectomy. Subjects must be smoke free and have not taken regular yoga classes 6 months prior to enrollment. Subjects will participate in twice weekly yoga sessions for 8 weeks and complete 4 quality of life forms 5 times during study.

DETAILED DESCRIPTION:
The feasibility study refers to the ability to recruit patients willing to participate in the Eischens yoga interventional arm. Those who are recruited during the feasibility study are seemlessly move to the Phase II study, and for this reason the feasibility study and Eischens yoga interventional arms are reported simply as the Eischens yoga interventional arm.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Prostate cancer patients undergoing active radiation therapy (external beam radiation with photons and/ or protons). Prior or concurrent androgen deprivation therapy is permitted.
* Patients of age >18 years, and all races will be included in the study.
* Patients must have an ECOG Performance Score ≤ 1
* All patients must sign an informed consent form

Caregivers

* Subject is age >18 years
* Subject is English-speaking
* Subject must sign an informed consent form

Exclusion Criteria

Patients

* Patients with medical restrictions that may interfere with or prevent them from taking part in the yoga interventions per their physician orders as evaluated by ECOG Performance Status score.
* Active, regular cigarette smokers, such that smoking may interfere with relaxation and breathing modalities of the yoga interventions. (Smokers that have been smoke-free for 6 months may be included)
* Patients who currently practice or have recently practiced yoga (taken a yoga class on a regular basis in the last 6 months).
* Patients who are undergoing chemotherapy for any reason
* Patients with evidence of metastatic disease

Caregivers

* Subjects that are unwilling or unable to provide informed consent
* Subjects with medical restrictions that may interfere with or prevent them from taking part in the yoga interventions
* Active, regular cigarette smokers, such that smoking may interfere with relaxation and breathing modalities of the yoga interventions. (Smokers that have been smoke-free for 6 months may be included)
* Patients who currently practice or have recently practiced yoga (taken a yoga class on a regular basis in the last 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with stage I or II prostate cancer undergoing radiation therapy. Enrolled subjects will not have smoked nor taken any regular yoga classes in the 6 months preceding their participation in the study.
  Additionally they will have not undergone a surgical prostatectomy
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neha Vapiwala, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Feasibility Phase and Phase II: Radiotherapy and Eischens Yoga have been combined because the feasibility phase's purpose was to identify and recruit patients willing to participate in the Phase II: Radiotherapy and Eischens Yoga. Those in the feasibility are seamlessly enrolled in the Phase II: Radiotherapy and Eischens Yoga.
Groups:
- Feasibility/Phase II: Radiotherapy and Eischens Yoga: Radiotherapy and Eischens Yoga
- Phase II: Radiotherapy Without Eischens Yoga: Radiotherapy without Eischens Yoga
Period: Overall Study
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Without Eischens Yoga
Started | 35 | 33
Completed | 22 | 28
Not Completed | 13 | 5

BASELINE CHARACTERISTICS:
Population: Feasibility Phase and Phase II: Radiotherapy and Eischens Yoga have been combined because the feasibility phase's purpose was to identify and recruit patients willing to participate in the Phase II: Radiotherapy and Eischens Yoga. Those in the feasibility are seamlessly enrolled in the Phase II: Radiotherapy and Eischens Yoga
Groups:
- Total: Total of all reporting groups
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Without Eischens Yoga | Total
Number analyzed (Participants) | 22 | 28 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 17 | 23 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (6.7) | 72.8 (7.0) | 72.08 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 28 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 28 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 19 | 24 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 22 | 28 | 50

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Time Frame: 8 weeks
Measure: Number; unit: Adverse Events
Groups:
- Feasibility/Phase II: Radiotherapy and Eischens Yoga: Radiotherapy with Eischens Yoga
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Without Eischens Yoga
Number analyzed (Participants) | 22 | 28
Adverse Events | 0 | 0

2. Secondary Outcome: Brief Fatigue Inventory Score
Description: A 9 item 11 point Likert-scale that rapidly assesses fatigue severity 0 - 90 range with greater numbers indicating greater levels of fatigue
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Phase II: Radiotherapy Without Eischens Yoga: Radiotherapy
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Without Eischens Yoga
Number analyzed (Participants) | 22 | 28
score on a scale | 12.2 (16.3) | 27.4 (18.3)

3. Secondary Outcome: Functional Assessment of Cancer Therapy: Physical Well-Being Score
Description: 7 item 5 point Likert-scale questionnaire. 0 - 35 range with larger number implies better physical well-being
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Without Eischens Yoga
Number analyzed (Participants) | 22 | 28
score on a scale | 24.9 (2.3) | 24.3 (3.0)

4. Secondary Outcome: Functional Assessment of Cancer Therapy: Social Well-Being Score
Description: 7 item 5 point Likert-scale questionnaire. 0 - 35 range with larger number implies better social well-being
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Without Eischens Yoga
Number analyzed (Participants) | 22 | 28
score on a scale | 23.5 (2.1) | 21.4 (3.6)

5. Secondary Outcome: Functional Assessment of Cancer Therapy: Emotional Well-Being Score
Description: 6 item 5 point Likert-scale questionnaire. 0 - 30 range with larger number implies better emotional well-being
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Without Eischens Yoga
Number analyzed (Participants) | 22 | 28
score on a scale | 20.1 (3.4) | 21.0 (2.2)

6. Secondary Outcome: Functional Assessment of Cancer Therapy: Functional Well-Being
Description: 7 item 5 point Likert-scale questionnaire. 0 - 35 range with larger number implies better functional well-being
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Without Eischens Yoga
Number analyzed (Participants) | 22 | 28
score on a scale | 22.5 (4.8) | 21.4 (4.0)

7. Secondary Outcome: International Index of Erectile Function Score
Description: 5 item and 5 point Likert-scale The scores range from 0 to 25, with scores >21 indicating normal erectile function and scores <12 indicating moderate to severe ED
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Without Eischens Yoga
Number analyzed (Participants) | 22 | 28
score on a scale | 22.5 (4.8) | 21.4 (4.0)

8. Secondary Outcome: International Prostate Symptom Score
Description: 8 item 6 point Likert-scale Scores on this scale range from 0 to 35, with a score of 8 to 19 indicating moderate urinary symptoms and 20 to 35 severe urinary symptoms
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Without Eischens Yoga
Number analyzed (Participants) | 22 | 28
score on a scale | 10.8 (8.1) | 15 (6.4)

ADVERSE EVENTS:
Time Frame: 8 Weeks
Description: Feasibility Phase and Phase II: Yoga Group have been combined because the feasibility phase's purpose was to identify and recruit patients willing to participate in the Phase II: Yoga Group. Those in the feasibility are seamlessly enrolled in the Phase II: Yoga Group.
Groups:
- Phase II: Radiotherapy Wihtout Eischens Yoga: Radiotherapy without Eischens Yoga
Arm/Group | Feasibility/Phase II: Radiotherapy and Eischens Yoga | Phase II: Radiotherapy Wihtout Eischens Yoga
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/28
Other Adverse Events (participants affected / at risk) | 0/22 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT02135653/Prot_SAP_000.pdf